CLINICAL TRIAL: NCT03373292
Title: Evaluation of the Feasibility, Safety and Efficacy of Venous Stenting for Internal Jugular Vein Stenosis
Brief Title: Endovascular Stenting Treatment for Patients With Internal Jugular Vein Stenosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, Vice President, Professor, Xuanwu Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stenting2018-IJVS
Record Dates: First submitted 2017-12-03; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Stent Stenosis; Intracranial Hypertension; Headache; Tinnitus; Papilledema; Visual Impairment
Keywords: Stenting; Jugular vein stenosis; Intracranial hypertension; Headache; Tinnitus; Papilledema; Visual impairment
MeSH Terms: conditions — Intracranial Hypertension; Headache; Tinnitus; Papilledema; Vision Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venous stenting (Group-1) (Experimental): Patients in this group will undergo venous stenting treatment at once after enrollment.
  Interventions: Procedure: Venous stenting for internal jugular vein stenosis
- Stenting one-month after routine medical treatment (Group-2) (Experimental): Patients in this group will undergo routine medical treatment for one month, followed by venous stenting intervention.
  Interventions: Procedure: One-month routine medical treatment followed by venous stenting for internal jugular vein stenosis

INTERVENTIONS:
Procedure: Venous stenting for internal jugular vein stenosis — After confirming the diagnosis of IJVS by Jugular Vein Doppler Ultrasound, Magnetic Resonance Venography (MRV) and/or Computed Tomography Venography (CTV), and excluding external compression-induced stenosis as well as other causes of intracranial pressure elevation, patients will be divided into two groups randomly (30 for each group: group-1 and group-2).
  Patients in Group-1 will receive Digital Subtraction Angiography (DSA) immediately after enrollment, and trans-stenotic pressures (∆MPGs) will be measured, balloon angioplasty bridging venous stenting will be performed when their ∆MPGs of jugular veins are equal to or greater than 5.44 cmH₂O (4 mmHg).
  Arms: Venous stenting (Group-1)
Procedure: One-month routine medical treatment followed by venous stenting for internal jugular vein stenosis — Patients in Group-2 will receive routine medical treatment for one month. Afterwards, they will undergo DSA (the procedure is the same as that in Group-1).
  Notably, patients in Group-2 with medical uncontrolled intracranial hypertension will be provided stenting of their jugular veins at any time during the one-month routine medical treatment, in attempt to reduce their intracranial pressure and ameliorate visual damages in time.
  Arms: Stenting one-month after routine medical treatment (Group-2)

SUMMARY:
This is a prospective, randomized, single-center clinical study aiming to explore the safety and efficacy of venous stenting for patients with internal jugular vein stenosis (IJVS).

DETAILED DESCRIPTION:
The role of isolated non-thrombotic IJVS in idiopathic intracranial hypertension has recently gained a vested interest. Compared with venous sinus stenosis, isolated IJVS at extracranial segments is more concealed and likely to be neglected, leading to misdiagnosis or treatment delay and subsequent exacerbation of clinical outcomes. Stenting seems to hold a potential of addressing the intracranial pressure elevation-associated clinical issues from etiological level, especially after medical therapy failure. The complications of stenting such as ipsilateral headache, restenosis, intra-stent thrombosis and hemorrhage have beem demonstrated in the settings of intracranial sinus obstruction and osseous impingement-associated IJVS, particularly bony structures between the styloid process and lateral mass of C1 that constrain the IJV. Nevertheless, so far, to the best of our knowledge, few or no stenting related adverse events have been found in isolated IJVS patients with venous stent implantation.

In this study, 60 patients satisfied with the inclusion criteria will be enrolled and randomly allocated into two groups. The safety and efficacy of stenting in patients with non-osseous impingement-mediated IJVS will be analyzed. Other medical interventions will be guaranteed according to the best medical judgment from clinical practitioners.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 to 80 years of age, both genders.
2. Patients diagnosed with IJVS surrounded by abnormally and tortuous collateral veins verified by MRV, CTV and/or DSA.
3. Pressure gradient across the stenotic segments is equal to or greater than 4 mmHg.
4. Intracranial hypertension associated manifestations cannot be satisfactorily controlled by conservative or non-surgical therapies.
5. Informed consent obtained from the patient or his/her health care proxy, able to cooperate follow-up visits.

Exclusion Criteria:

1. External osseous impingement associated IJVS.
2. Contraindication to iodinated contrasts.
3. Contraindication to general anesthesia.
4. Contraindication to standard medical therapy such as Aspirin, Clopidogrel or anticoagulants.
5. Intracranial abnormalities such as tumor, abscess, vascular malformation, cerebral venous sinus stenosis or thrombosis.
6. Previous history of major surgeries within 30 days prior to inclusion, or scheduled for any of the procedures within 12 months after inclusion.
7. Severe hematological, hepatic or renal dysfunctions.
8. Current or having a history of chronic physical diseases or mental disorders.
9. Pregnant or lactating women.
10. Life expectancy < 1 year due to concomitant life-threatening illness.
11. Patients unlikely to be compliant with intervention or return for follow-up visits.
12. No signed consent from the patient or available legally authorized representatives.
13. Patients recruited to other clinical trials with medications or devices, which may affect the outcome of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Correction of internal jugular vein stenosis (IJVS) and abnormal collateral veins | baseline, 1, 6 and 12 months
  The status of internal jugular vein blood flow and collateral veins will be evaluated by imaging modalities, mainly including: Jugular Vein Doppler Ultrasound, Magnetic Resonance Venography (MRV), Computed Tomography Venography (CTV) and Digital Subtraction Angiography (DSA).

SECONDARY OUTCOMES:
The evaluation of cerebral spinal fluid (CSF) pressure | baseline, immediately post-stenting, within 1 month
  CSF pressure will be assessed by lumbar puncture.
The evaluation of headache | baseline, within 1, 6 and 12 months
  The intensity of headache will be assessed with the Headache Impact Test-6 (HIT-6).
The evaluation of tinnitus | baseline, within 1, 6 and 12 months
  The severity of tinnitus will be assessed by the Tinnitus Handicap Inventory Questionnaire (THIQ).
The evaluation of the severity of papilledema and other ophthalmological conditions | baseline, within 1, 6 and 12 months
  The severity of papilledema will be assessed based on Frisén papilledema grade (FPG) criteria; the assessment of other ophthalmological conditions including visual acuity, visual ﬁeld, and fundus etc. will be based on visual acuity chart, visual fields picture, and optical coherence tomography (OCT) etc.
Changes in cerebral white matter (WM) | baseline, within 12 months
  The characteristics of WM will be evaluated by Magnetic Resonance Imaging (MRI).
The evaluation of cognitive function | baseline, within 12 months
  Cognitive function will be assessed with the Mini-Mental State Examination (MMSE), the Montreal Cognitive Assessment (MoCA) and/or the Modified Telephone Interview for Cognitive Status (TICS-M).
The evaluation of mental status | baseline, within 12 months
  Mental status will be assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS score ranges between 0 and 21 for either anxiety or depression. A cut-off point of 8/21 is indicated for anxiety or depression.
The evaluation of sleeping status | baseline, within 12 months
  Sleeping status will be assessed with the Pittsburgh Sleep Quality Index (PSQI) and/or the Athens Insomnia Scale (AIS). The PSQI score provides an overall score ranging from 0 to 21, where a cut-off score of ≤5 denotes a healthier sleep quality. The AIS score provides an overall score ranging from 0 to 24, where a cut-off score of <6 denotes a healthier sleep quality.
The extent of disability or dependence in the daily activities | baseline, within 12 months
  The extent of disability will be assessed by the modified Rankin Scale (mRS). (Score 0-no symptoms; score 1-no significant disability; score 2-slight disability; score 3-moderate disability; score 4-moderately severe disability; score 5-severe disability; score 6-dead.)
Percentage of participants with abnormal lab values | baseline, within 12 months
  Lab examinations such as hepatic and renal function, blood and urine routine will be recorded.
Percentage of participants with procedure-related and/or stenting-related complications | within 12 months
The incidence of all cause mortality | within 12 months
  Death secondary to any reasons

CONTACTS AND LOCATIONS:
Overall Officials: Xuming Ji, MD, PhD, Study Director — Xuanwu Hosptial, Capital Medical University; Ran Meng, MD, PhD, Principal Investigator — Xuanwu Hosptial, Capital Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou D, Meng R, Zhang X, Guo L, Li S, Wu W, Duan J, Song H, Ding Y, Ji X. Intracranial hypertension induced by internal jugular vein stenosis can be resolved by stenting. Eur J Neurol. 2018 Feb;25(2):365-e13. doi: 10.1111/ene.13512. Epub 2017 Dec 7. PMID 29114973
- [Background] Higgins JN, Garnett MR, Pickard JD, Axon PR. An Evaluation of Styloidectomy as an Adjunct or Alternative to Jugular Stenting in Idiopathic Intracranial Hypertension and Disturbances of Cranial Venous Outflow. J Neurol Surg B Skull Base. 2017 Apr;78(2):158-163. doi: 10.1055/s-0036-1594238. Epub 2016 Nov 23. PMID 28321380
- [Background] Spitze A, Malik A, Lee AG. Surgical and endovascular interventions in idiopathic intracranial hypertension. Curr Opin Neurol. 2014 Feb;27(1):69-74. doi: 10.1097/WCO.0000000000000049. PMID 24296639
- [Derived] Ding J, Liu Y, Li X, Chen Z, Guan J, Jin K, Wang Z, Ding Y, Ji X, Meng R. Normobaric Oxygen May Ameliorate Cerebral Venous Outflow Disturbance-Related Neurological Symptoms. Front Neurol. 2020 Nov 13;11:599985. doi: 10.3389/fneur.2020.599985. eCollection 2020. PMID 33281736